CLINICAL TRIAL: NCT01460511
Title: Phase III Study of Epinephrine Inhalation Aerosol for Evaluation of Efficacy and Safety of E004 in Children With Asthma
Brief Title: Evaluation of Efficacy and Safety of E004 in Children With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: API-E004-CL-D
Record Dates: First submitted 2011-10-24; First posted 2011-10-27 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Asthma
Keywords: Mild bronchial asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- P - Placebo-HFA (Placebo Comparator): Placebo-HFA, 0 mcg/inhalation, 2 inhalations QID
  Interventions: Drug: Placebo-HFA
- T - E004 (Epinephrine Inhalation Aerosol) HFA-MDI (Experimental): E004 (Epinephrine Inhalation Aerosol) HFA-MDI, 125 mcg/inhalation, 2 inhalations QID
  Interventions: Drug: E004 (Epinephrine Inhalation Aerosol) HFA-MDI

INTERVENTIONS:
Drug: E004 (Epinephrine Inhalation Aerosol) HFA-MDI — E004 (Epinephrine Inhalation Aerosol) HFA-MDI, 125 mcg/inhalation, 2 inhalations QID
  Arms: T - E004 (Epinephrine Inhalation Aerosol) HFA-MDI
Drug: Placebo-HFA — Placebo-HFA, 0 mcg/inhalation, 2 inhalations QID
  Arms: P - Placebo-HFA

SUMMARY:
This is a multi-center, randomized, double-blinded, placebo-controlled, parallel, 4-week study in 60 pediatric patients (4-11 years old) with asthma, comparing E004 with Placebo HFA-MDI in pediatric patients who are 4-11 years of age with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy male, and premenarchal female, children aged 4 - 11 years upon Screening.
* With documented asthma, requiring inhaled epinephrine or beta2-agonist treatment, with or without concurrent anti-inflammatory therapies for at least 6-months prior to Screening.
* Being capable of performing spirometry for FEV1
* Satisfying criteria of asthma
* Can tolerate withholding treatment with inhaled bronchodilators and other allowed medications for the minimum washout periods
* Demonstrating a Screening Baseline FEV1 that is 50 - 90% of Polgar predicted normal value.
* Demonstrating an Airway Reversibility,
* Demonstrating satisfactory techniques in the use of a metered-dose inhaler (MDIs) and a hand held peak expiratory flow meter, after training.
* Has been properly consented to participate in this study.

Exclusion Criteria:

* Any current or past medical conditions that, per investigator discretion, might significantly affect pharmacodynamic responses to the study drugs
* Concurrent clinically significant cardiovascular, hematological, renal, neurologic, hepatic, endocrine, psychiatric, or malignant diseases.
* Known intolerance or hypersensitivity to any component of the study drugs
* Recent infection of the respiratory tract
* Use of prohibited medications
* Having been on other investigational drug/device studies in the last 30 days prior to screening.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint AUC of FEV1's relative change | Visit 1 and Visit 3 at 5, 30, 60, 120, 180, 240, and 360 minutes post-dose
  bronchodilator effect expressed as AUC of FEV1's relative change (from the same day baseline) versus time, defined as AUC of ΔFEV1%.

SECONDARY OUTCOMES:
AUC of FEV1 volume changes (AUC of change in FEV1) | Visit 1 and Visit 3 at 5, 30, 60, 120, 180, 240, and 360 minutes post-dose
  determination of the change in FEV1 from baseline at visit to to post treatment at Visit 3
Maximum of change in FEV1% (Fmax) | Visit 1 and Visit 3 at 5, 30, 60, 120, 180, 240, and 360 minutes post-dose
  Evaluation of maximum percent change in FEV1
Curves of change in FEV1, and change in FEV1%, versus time | Visit 1 and Visit 3 at 5, 30, 60, 120, 180, 240, and 360 minutes post-dose
  Evaluation of curves of change in FEV1 and percent change in FEV1 over time
Time to onset of bronchodilator effect (to onset), determined the time point (within 60 minutes) where FEV1 first reaches ≥12% above Same-Day Baseline. | Study Visits 1and 3 within 60 minutes post dose
  Evaluation of how much time elapses (within 60 minutes), until FEV1 first reaches ≥12% above Same-Day Baseline.
The time to peak FEV1 effect (tmax), defined as the time of Fmax. | Study Visits 1 and 3 at 5, 30, 60, 120, 180, 240, and 360 minutes post-dose
  Evaluation of how much time elapses until FEV1 reaches its peak
Duration of efficacy (duration), defined as the total length of time when ΔFEV1% reaches and stays ≥12% above Same-Day Baseline. | Study Weeks 1and 3 at 5, 30, 60, 120, 180, 240, and 360 minutes post-dose
  Evaluation of the total length of time it takes until the change in FEV1% reaches and stays ≥12% above Same-Day Baseline.
Percentage of positive responders (R%), including all subjects whose Fmax reaches ≥12% above Same-Day Baseline. | Study Weeks 1 and 3 within 60 minutes post dose
  Evaluation of what percentage of subjects are positive responders (R%), including all subjects whose Fmaxreaches ≥12% above Same-Day Baseline.
Mean daily morning pre-dose Peak Expiratory Flow Rate (PEF) | daily pre-dose
  Evaluation of the mean of daily morning pre-dose Expiratory Flow Rate
Evaluation of Vital Signs | predose, and 3, 20, 60, 360 minutes post-dose
  Monitoring of vital signs (SBP/DBP, and heart rate) at the Screening Visit (Baseline and 30 min post-dose), and at the baseline, 3, 20, 60 and 360 minute time points during the study
12-lead ECG | Pre-dose and , 3, 20 and 60 minutes post-dose (Study Visits 1 and 3)
  Recording of 12-lead ECG (Routine and QT/QTc) at Screening Visit Baseline, and at the baseline, 3, 20 and 60 minute time points during Study Visits 1 and 3
Albuterol HFA usage for rescue relief of acute asthma symptoms | Study Visits 1, 2, and 3, within 30 min predose
  Evaluation Albuterol HFA usage for rescue relief of acute asthma symptoms

CONTACTS AND LOCATIONS:
Overall Officials: John Gao, M.D., Study Chair — Amphastar Pharmaceuticals, Inc.
Locations (8):
- United States (8):
  - Amphastar Site 5, Costa Mesa, California
  - Amphastar Site 8, Orange, California
  - Amphastar Site 4, Stockton, California
  - Amphastar Site 2, Medford, Oregon
  - Amphastar Site 1, Portland, Oregon
  - Amphastar Site 7, North Charleston, South Carolina
  - Amphastar Site 3, El Paso, Texas
  - Amphastar Site 6, San Antonio, Texas

REFERENCES:
- [Background] Pinnas JL, Schachtel BP, Chen TM, Roseberry HR, Thoden WR. Inhaled epinephrine and oral theophylline-ephedrine in the treatment of asthma. J Clin Pharmacol. 1991 Mar;31(3):243-7. doi: 10.1002/j.1552-4604.1991.tb04969.x. PMID 2019665
- [Background] Hendeles L, Marshik PL, Ahrens R, Kifle Y, Shuster J. Response to nonprescription epinephrine inhaler during nocturnal asthma. Ann Allergy Asthma Immunol. 2005 Dec;95(6):530-4. doi: 10.1016/S1081-1206(10)61014-9. PMID 16400891
- [Background] Warren JB, Doble N, Dalton N, Ewan PW. Systemic absorption of inhaled epinephrine. Clin Pharmacol Ther. 1986 Dec;40(6):673-8. doi: 10.1038/clpt.1986.243. PMID 3780129
- [Background] Cripps A, Riebe M, Schulze M, Woodhouse R. Pharmaceutical transition to non-CFC pressurized metered dose inhalers. Respir Med. 2000 Jun;94 Suppl B:S3-9. PMID 10919679
- [Background] Dickinson BD, Altman RD, Deitchman SD, Champion HC. Safety of over-the-counter inhalers for asthma: report of the council on scientific affairs. Chest. 2000 Aug;118(2):522-6. doi: 10.1378/chest.118.2.522. PMID 10936150